CLINICAL TRIAL: NCT04207957
Title: A Phase I, Open-label, Randomised Biopharmaceutics Study in Healthy Subjects to Evaluate the Pharmacokinetics, Safety and Tolerability of Single Doses of IV and Oral Formulations of Olorofim
Brief Title: A Biopharmaceutics Study to Assess the Pharmacokinetics of Single Oral and IV Doses of Olorofim
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: F901318-01-14
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Intervention Model Description: 3 Treatment Periods for Cohorts A and B 2 Treatment Periods for Cohort C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IV (Other): 2 h IV infusion (Groups A/B)
  Interventions: Drug: Olorofim
- oral (fasted) (Other): 30 mg tablets given after an overnight fast (Groups A/B)
  Interventions: Drug: Olorofim
- oral (fed) (Other): 30 mg tablets given after a high fat breakfast (Groups A/B)
  Interventions: Drug: Olorofim
- oral (intact tablet) (Other): 30 mg tablets (Group C)
  Interventions: Drug: Olorofim
- oral (NG tube) (Other): 30 mg tablets in water via NG tube (Group C)
  Interventions: Drug: Olorofim

INTERVENTIONS:
Drug: Olorofim — 150 mg
  Other Names: F901318

SUMMARY:
This is a Phase I, single-centre, randomised, open-label, crossover study in 24 healthy subjects. Twelve subjects will each receive olorofim as a single IV infusion, single oral dose (fasted) and single oral dose (fed) and 12 subjects will each receive olorofim orally as intact tablets and via NG tube

ELIGIBILITY:
Inclusion Criteria:

* males or females of any ethnic origin between 18 and 55 years of age
* subjects weighing between 50 and 100 kg, with a body mass index (BMI) between 18 and 30 kg/m2.
* subjects in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations

Exclusion Criteria:

* Male subjects (or their partners) who are not willing to use appropriate contraception during the study and for 3 months after end of dosing.
* Female subjects who are pregnant or lactating.
* Subjects who have received any prescribed systemic or topical medication within 14 days of first dose administration
* Subjects who have used any non-prescribed systemic or topical medication within 7 days of first dose administration
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of first dose administration
* Subjects with or history of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatry, respiratory, metabolic, endocrine, ocular haematological or other major disorders as determined by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) for olorofim | 35 days
area under the concentration time curve to time of last quantifiable concentration (AUC0-tlast) for olorofim | 35 days
Absolute bioavailability of olorofim (F) | 35 days

SECONDARY OUTCOMES:
Time to Cmax (TMax) for olorofim | 35 days
area under the concentration time curve to infinity (AUC0-∞) for olorofim | 35 days
terminal elimination half-life (t½) for olorofim | 35 days
Number of subjects with treatment-related adverse events | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, Principal Investigator — Covance CRU
Locations (1):
- Covance Clinical Research Unit, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No